CLINICAL TRIAL: NCT02918539
Title: Registry of Amyloid Positive Patients for Alzheimer's Disease Drug Research Trials
Acronym: RAmP
Status: Completed | Type: Observational
Sponsor: Avid Radiopharmaceuticals (Industry)
Collaborators: Eli Lilly and Company (Industry); PRA Health Sciences (Industry)
Responsible Party: Sponsor
Other Study IDs: 18F-AV-45-A25; PRA Study Code: 446601 (Other: PRA Health Sciences)
Record Dates: First submitted 2016-09-13; First posted 2016-09-29 (Estimated); Last update posted 2018-10-24 (Actual); Status verified 2018-10

CONDITIONS: Alzheimer Disease; Cognition Disorders
MeSH Terms: conditions — Alzheimer Disease; Cognition Disorders | interventions — florbetapir

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- RAmP Registry Patients: Patients who have a) objectively verified cognitive impairment and etiology diagnosed or suspected to be Alzheimer's disease and b) a positive amyloid scan from either an existing amyloid scan that has been interpreted as positive or a florbetapir F 18 PET scan via protocol addendum
  Interventions: Drug: florbetapir F 18 PET scan

INTERVENTIONS:
Drug: florbetapir F 18 PET scan — For those patients who do not have an existing amyloid scan, each will receive an IV injection, 370 MBq (10 mCi), single dose of florbetapir F 18 followed by a Positron Emission Tomography (PET) Scan to determine amyloid status
  Other Names: Amyvid

SUMMARY:
This registry will be used to identify patients who have etiology diagnosed or suspected to be Alzheimer's disease and positive amyloid scans, and have indicated their interest in being contacted for an Eli Lilly and Company (Lilly) Alzheimer's Disease drug research trial.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients ≥ 50 years of age at the time of consent;
* Patients who have objectively verified cognitive impairment and etiology diagnosed or suspected to be Alzheimer's disease;
* Patients who are willing to make available to Avid a positive amyloid scan, or if an amyloid scan is not available, are willing to undergo amyloid scanning via the Florbetapir F 18 PET Scan Addendum;
* Patients who are willing to be contacted for possible participation in Lilly drug research trials targeting Alzheimer's disease;
* Patients who give informed consent or have a legally authorized representative (LAR) to consent for enrollment; and
* Patients who have a partner (informant) who is willing to participate as a source of information and has at least weekly contact with the patient (contact can be inperson, via telephone or electronic communication). The informant must have sufficient contact such that the referring physician feels the informant can provide meaningful information about the patient.

Exclusion Criteria:

* Patients who have a Mini Mental State Examination (MMSE) score of < 16;
* Patients who have an amyloid-negative PET scan (either a historical scan or scan via the Florbetapir F 18 PET Scan Addendum);
* Patients who have serious or unstable medical conditions that would exclude completion of all procedures and data collection for the registry, or would be likely to preclude participation in a drug research trial;
* Patients who are currently participating in a clinical trial with an investigational agent; or
* Patients who, in the opinion of the physician, are otherwise unsuitable for this registry.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have a) objectively verified cognitive impairment and etiology diagnosed or suspected to be Alzheimer's disease and b) a willingness to make available to Avid a preexisting amyloid scan that has been interpreted as positive, or if an amyloid scan is not available, a willingness to undergo amyloid scanning via the Florbetapir F 18 PET Scan Addendum, will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 317 (Actual)
Dates: Start 2016-10; Primary Completion 2017-10-18 (Actual); Study Completion 2017-10-18 (Actual)

PRIMARY OUTCOMES:
Patient Registry Participation | Two years
  There is no formal hypothesis to test in this registry study. The registry will collect contact information of amyloid positive patients with cognitive impairment who have indicated interest in being contacted for a Lilly AD drug research trial. The primary outcome measure to be reported is the total number of participants in the registry.

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Chair — Avid Radiopharmaceuticals, Inc.
Locations (75):
- United States (75):
  - Arrowhead Internal Medicine, PC, Glendale, Arizona
  - Center for Neuro and Spine Inc. (CNS) - Main Office, Phoenix, Arizona
  - Imaging Endpoints, Scottsdale, Arizona
  - Center for Neurology and Spine, Sun City, Arizona
  - Woodland Research Northwest, Rogers, Arkansas
  - Neurology Center of North Orange County, Fullerton, California
  - Irvine Center for Clinical Research, Irvine, California
  - Senior Clinical Trials, Inc., Laguna Hills, California
  - Pacific Research Network, San Diego, California
  - Syrentis Clinical Research, Santa Ana, California
  - North Bay Neuroscience Institute, Sebastopol, California
  - Mile High Research Center, Denver, Colorado
  - Coastal Conneticut Research, New London, Connecticut
  - JEM Research Institute, Atlantis, Florida
  - Ptak Alzheimer Research Center, Clearwater, Florida
  - Wisdom Clinical Research Institute, Coral Gables, Florida
  - Direct Helpers Research, Hialeah, Florida
  - Healing Touch C&C Research Inc, Hialeah, Florida
  - Galiz Research, Hialeah, Florida
  - Advanced Research Institute of Miami, Homestead, Florida
  - Precision Clinical Research, Lauderdale Lakes, Florida
  - Neurology Associates, PA, Maitland, Florida
  - Merritt Island Medical Research, Merritt Island, Florida
  - Homestead Associates in Research, Miami, Florida
  - Dade Research Center, Miami, Florida
  - United Clinical Research, Corp., Miami, Florida
  - Advanced Medical Research Institute (AMRI), Miami, Florida
  - New Horizon Research Center, Miami, Florida
  - Advance Research Development Solutions, Miami Lakes, Florida
  - Bravo Health Care Center, North Bay Village, Florida
  - Laszlo J. Mate, MD, North Palm Beach, Florida
  - Pines Care Research Center, Pembroke Pines, Florida
  - Neurostudies.net, LLC, Port Charlotte, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Suncoast Neuroscience Associates, Inc., St. Petersburg, Florida
  - Olympian Clinical Research - South Tampa Office, Tampa, Florida
  - Tampa Neurology Associates, Tampa, Florida
  - University of South Florida Health Byrd Alzheimer's Institute, Tampa, Florida
  - Lovelance Scientific Resources, Inc., Venice, Florida
  - Sand Lake Imaging, MRI Facility, Winter Park, Florida
  - Doctors Clinical Research, Atlanta, Georgia
  - iResearch Atlanta, Decatur, Georgia
  - Community Hospital of Anderson and Madison Country, Anderson, Indiana
  - American Health Network of Indiana, Avon, Indiana
  - American Health Network of Indiana, LLC, Franklin, Indiana
  - Cotton O'Neil Clinical Research Center, Topeka, Kansas
  - Sheppard Pratt Health System, Baltimore, Maryland
  - Spectrum Clinical Research, Baltimore, Maryland
  - Boston Center for Memory, Brookline, Massachusetts
  - Michigan State University, East Lansing, Michigan
  - Hattiesburg Clinic, Hattiesburg, Mississippi
  - Millenium Psychiatric Associates, Creve Coeur, Missouri
  - Las Vegas Medical Center, Las Vegas, Nevada
  - Amici Clinical Research, Martinsville, New Jersey
  - The Cognitive and Research Center of New Jersey, Springfield, New Jersey
  - Advanced Memory Research Institute of NJ, PC, Toms River, New Jersey
  - Neurology Specialists of Monmouth County, PA, West Long Branch, New Jersey
  - Integrative Clinical Trials, Brooklyn, New York
  - Adirondack Medical Research, Glens Falls, New York
  - Neurological Associates of Long Island, Lake Success, New York
  - Richmond Behavioral Associates, Staten Island, New York
  - Dayton Center for Neurological Disorders, Dayton, Ohio
  - Clinical Inquest Center, Dublin, Ohio
  - Tulsa Clinical Research, LLC, Tulsa, Oklahoma
  - Legacy Research Institute, Portland, Oregon
  - Adler Institute for Advanced Imaging, Jenkintown, Pennsylvania
  - Pearl Clinical Research, Norristown, Pennsylvania
  - Rhode Island Mood and Memory Research Institute, East Providence, Rhode Island
  - Heights Doctors Clinic, Houston, Texas
  - Yvonne Kew MD PLLC Neuro-Oncology Clinic, Houston, Texas
  - FMC Science, Lampasas, Texas
  - The Clinical Research Group, Inc., Lewisville, Texas
  - Texas Medical Research Associates, LLC, San Antonio, Texas
  - National Clinical Research-Richmond, Inc., Richmond, Virginia
  - Dean Foundation for Health, Research and Education, Inc., Middleton, Wisconsin